CLINICAL TRIAL: NCT02855242
Title: Gut Microbiota Changes in Obese Individuals Undergoing Dedicated Lifestyle Modification Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Purna C. Kashyap, MBBS, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-001912
Record Dates: First submitted 2016-06-21; First posted 2016-08-04 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Program Group (Other): Lifestyle Counseling
  Interventions: Behavioral: Lifestyle Counseling
- Controls Group (Active Comparator): No lifestyle counseling
  Interventions: Other: Controls Group

INTERVENTIONS:
Behavioral: Lifestyle Counseling — Participation in weekly group sessions over a period of 10 weeks, with information on healthy nutrition and exercises promoting weight loss
  Other Names: Obese group participants
  Arms: Intervention Program Group
Other: Controls Group — Subjects not participating in any lifestyle counseling
  Other Names: No Lifestyle Counseling
  Arms: Controls Group

SUMMARY:
The human gut microbiota has become the subject of extensive research in recent years, particularly in regards to the role it plays in obesity. Although lifestyle factors, diet, and lack of exercise contribute largely to this obesity epidemic, there is increasing evidence that the human gut microbiota also influences weight gain.

The investigators hope to learn more information about the change in gut microbiota, especially with regards to those who are successful with weight loss, versus those who don't lose weight, after participating in a lifestyle modification program at the Dan Abraham Healthy Living Center (DAHLC).

DETAILED DESCRIPTION:
The gut microbiome is altered in obesity and is being increasingly studied given its role in energy harvest and fat storage with the hopeful goal of discovering a modifiable intervention to affect obesity and its consequences. Mouse models have already shown that transplantation of an obese microbiota into germ-free mice yields increased adiposity compared to transplantation of a lean microbiota. In humans, initial studies looked at the relative proportion of Bacteroidetes and Firmicutes in obese versus lean individuals and then followed those obese individuals who lost weight on low-calorie diets. The relative proportion of Bacteroidetes was decreased in obese people, and this then increased with weight loss. While certainly provocative, the findings were not consistently reproduced.

Subjects will include members of the Dan Abraham Healthy Living Center (DAHLC) program or the Healthy Living Program (HLP) at Mayo Clinic Rochester, who are seeking advice for weight management concerns.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and above;
* Subjects who are overweight or obese (BMI of 25 or greater);
* DAHLC/HLP eligible members who are able to access DAHLC support services;

Exclusion Criteria:

* Known diagnosis of inflammatory bowel disease, microscopic colitis, celiac disease or other inflammatory conditions;
* Antibiotic use within the past 4 weeks (they can be enrolled after a four week washout period and subsequent use during the 6 month study duration does not exclude them);
* Bowel preparation for colonoscopy within the past week;
* Pregnancy or plans to become pregnant within the study time frame;
* Vulnerable Adults;
* Any other disease(s), condition(s) or habit(s) that would interfere with completion of the study, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect study outcomes;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-04; Primary Completion 2020-07-28 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Changes in weight loss | baseline to 6 months
  enrolled in exercise program

SECONDARY OUTCOMES:
Changes in gut microbiota | Baseline to 6 months
  Gut microbiota, fecal metabolites will be identified using ultra performance liquid chromatography-mass spectrometry in the CTSA metabolomics core following extraction of fecal water samples

CONTACTS AND LOCATIONS:
Overall Officials: Purna C Kashyap, M.B.B.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared with Mayo Clinic research staff involved in this study; outside academic institutions, as specified in the protocol; and the Mayo Clinic Institutional Review Board that oversees the research.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials